CLINICAL TRIAL: NCT01498003
Title: Safety and Efficacy of Peri-procedural Use of Tirofiban in Elective Percutaneous Coronary Intervention for Long Coronary Lesions With Overlapping Drug-Eluting Stent
Brief Title: Tirofiban in Stenting for Long Coronary Lesion
Acronym: PETITION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhang Qi, MD, Vice Director of Cath. Lab, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20111211
Record Dates: First submitted 2011-12-11; First posted 2011-12-23 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease
Keywords: coronary disease; stents; thrombosis; myocardial infarction; prognosis
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Thrombosis; Myocardial Infarction | interventions — Tirofiban; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Placebo Comparator): normal saline was applied to those randomized to control group, with same use as tirofiban
  Interventions: Drug: normal saline solution
- Tirofiban group (Experimental): after angioram, and before guiding catheter engagement: 10μg/kg bolus followed by 0.15μg/kg/min maintenance infusion
  Interventions: Drug: tirofiban

INTERVENTIONS:
Drug: tirofiban — 10μg/kg bolus followed by 0.15μg/kg/min maintenance infusion for 12h
  Other Names: Xinweining, Grand Pharmaceutical Group, Wuhan, China
  Arms: Tirofiban group
Drug: normal saline solution — same use as tirofiban
  Arms: Control group

SUMMARY:
Periprocedural myonecrosis or infarction are associated with short, intermediate, and long term adverse outcomes. Previous study indicated 12.6% of patients suffered a peri-procedural CK-MB rise by overlapping use of drug-eluting stents for long coronary lesions. Here the investigators hypothesize that peri-procedural use of tirofiban could reduce the occurrence of periprocedural infarciton in elective patients with long coronary lesions treated by overlapping use of drug-eluting stents.

DETAILED DESCRIPTION:
According to the results of 12.6% occurrence of peri-procedural myocardial infarction after long stent implantation by previous report[International Journal of Cardiology 2009;134: 231-237], the investigator hypothesize the 50% reduction of peri-procedural MI by using tirofiban. Three hundred and sixty-nine patients in each group are needed to reach 80% of power with α 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18y~80y, with symptomatic coronary disease
* At least one lesion length more than 40mm to be treated by overlapping drug-eluting stents in major epicardial coronary vessel

Exclusion Criteria:

* Aspirin or clopidogrel intolerance
* Lesions length less than 40mm, or overlapping stent length less than 40mm
* Bifurcation lesions need to be treated by two stents
* Patients with acute coronary syndrome and elevated baseline cardiac enzyme (CK-MB)
* Left ventricular ejection fraction less than 0.35
* Baseline estimated GFR less than 30
* Estimated life time less than one year
* Refuse to sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
periprocedural infarction | 12h after procedure
  definition of periprocedural MI is a CK elevation >3 times the upper limit of normal.

SECONDARY OUTCOMES:
major bleeding | during hospitalization (up to 2 weeks)
  The safety outcome of major bleeding according to the Thrombolysis in Myocardial Infarction (TIMI) definition
major adverse cardiac event | one year after procedure
  major adverse cardiac event (MACE) includes cardiac death, target vessel revascularization, and re-occurrence of myocardial infarction after discharge

CONTACTS AND LOCATIONS:
Overall Officials: WeiFeng Shen, PhD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang Q, Wang XL, Liao ML, Hu J, Yang ZK, Ding FH, Zhang JS, Du R, Zhu TQ, Shen WF, Zhang RY. Periprocedural use of tirofiban in elective percutaneous coronary intervention for long coronary lesions in stable patients with overlapping drug-eluting stents--the PETITION study: a prospective, randomized, multicenter study. Catheter Cardiovasc Interv. 2015 Mar;85 Suppl 1:762-9. doi: 10.1002/ccd.25864. PMID 25630513
- See also: published results — http://www.ncbi.nlm.nih.gov/pubmed/25630513